CLINICAL TRIAL: NCT01789593
Title: A Trial Investigating the Effect of Acute Hypoglycaemia on Cognitive Function and Brain Activation Patterns in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: NN1250-4001; U1111-1131-8749 (Other: WHO)
Record Dates: First submitted 2013-01-25; First posted 2013-02-12 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Glucose Clamp Technique

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypoglycaemia / euglycaemia clamp (Other)
  Interventions: Other: glucose clamp
- Euglycaemia clamp / hypoglycaemia (Other)
  Interventions: Other: glucose clamp

INTERVENTIONS:
Other: glucose clamp — Each subject will be randomly allocated to an experimental visit sequence consisting of a hypoglycaemic glucose clamp followed by euglycaemic glucose clamp (using i.v. infusion of human soluble insulin (Actrapid®)) or vice versa separated by at least 21 days. Each visit includes an overnight stay. For each of the two conditions (euglycaemia and hypoglycaemia) cognitive performance will be assessed by a validated cognitive test

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to compare cognitive function and associated brain activation patterns during an acute hypoglycaemic episode and during euglycaemia (normal blood glucose concentration). Additionally, the purpose is to assess cognitive function in the recovery phase after hypoglycaemia or euglycaemia, respectively, in subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed subjects
* Type 1 diabetes mellitus for at least 12 months
* Treated with multiple daily insulin injections or continuous subcutaneous insulin infusion (CSII) for at least 12 months
* Body mass index 18.0-28.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Current tobacco user (any smoking or use of nicotinic products within 3 months prior to screening)
* Visual impairment or auditory impairment

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2013-01-14 (Actual); Primary Completion 2013-12-01 (Actual); Study Completion 2013-12-01 (Actual)

PRIMARY OUTCOMES:
Digit Symbol Substitution Test (DSST) score | Average score during hypoglycaemia and/or euglycaemia measured 70-93 minutes after induction of hypoglycaemia and/or euglycaemia

SECONDARY OUTCOMES:
Regional cerebral blood flow (rCBF) score | Average score during hypoglycaemia and/or euglycaemia measured 70-93 minutes after induction of hypoglycaemia and/or euglycaemia
Paced Auditory Serial Addition Task (PASAT) score | During recovery from hypoglycaemia and/or euglycaemia measured 75-90 min after euglycaemia has been restored

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Århus C, Denmark

REFERENCES:
- [Result] Gejl M, Gjedde A, Brock B, Moller A, van Duinkerken E, Haahr HL, Hansen CT, Chu PL, Stender-Petersen KL, Rungby J. Effects of hypoglycaemia on working memory and regional cerebral blood flow in type 1 diabetes: a randomised, crossover trial. Diabetologia. 2018 Mar;61(3):551-561. doi: 10.1007/s00125-017-4502-1. Epub 2017 Nov 29. PMID 29188338
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com